CLINICAL TRIAL: NCT02222909
Title: Reverse Innovation and Patient Engagement to Improve Quality of Care and Patient Outcomes
Acronym: CONNECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CD-12-11-4948
Record Dates: First submitted 2014-08-18; First posted 2014-08-22 (Estimated); Results first posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2023-06

CONDITIONS: Diabetes; Cardiovascular Disease; Substance Abuse Disorder; Mental Health Disorder
Keywords: Community Based Organization; Reverse Innovation; Social Services; Referral; Chronic disease
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases; Substance-Related Disorders; Mental Disorders; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention CBOs (Experimental): Will receive "co-developed IT intervention" developed together with intervention group community based members. Set of primarily web based tools to improve connection with clients, Johns Hopkins Medicine and one another, referrals, and volunteer services.
  Interventions: Other: Co-developed IT intervention
- Control CBOs (No Intervention): Community Based Organizations that are being followed for data collection only for the period of one year

INTERVENTIONS:
Other: Co-developed IT intervention — The IT-based intervention is being co-developed with the community based organizations in the intervention group, and comprises tools to improve referral and tracking of clients, use of volunteers, and direct communication with hospital staff members
  Other Names: Healthify
  Arms: Intervention CBOs

SUMMARY:
Project CONNECT ("Community-based Organizations Neighborhood Network: Enhancing Capacity Together") is a randomized controlled trial that involves 22 community-based organizations (CBOs) located in Baltimore, MD. Half of these organizations were randomly assigned to the intervention group using a constrained cluster randomization process. The remaining 11 are a part of the control intervention group. The intervention is a co-developed set of IT tools hypothesized to improve the connections among intervention CBOs, Johns Hopkins health care facilities and CBO clients.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

Community Based Organization; 501-C3 status; Located within zip codes surrounding Johns Hopkins Hospital and Johns Hopkins Bayview Medical Center; Provides direct services to clients

Exclusion Criteria:

Part of Johns Hopkins Medicine or Baltimore City Agency

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6767 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert W Wu, MD MPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Zip codes surrounding Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD with other researchers.

REFERENCES:
- [Derived] Lowe D, Ryan R, Schonfeld L, Merner B, Walsh L, Graham-Wisener L, Hill S. Effects of consumers and health providers working in partnership on health services planning, delivery and evaluation. Cochrane Database Syst Rev. 2021 Sep 15;9(9):CD013373. doi: 10.1002/14651858.CD013373.pub2. PMID 34523117
- [Derived] Wu AW, Weston CM, Ibe CA, Ruberman CF, Bone L, Boonyasai RT, Hwang S, Gentry J, Purnell L, Lu Y, Liang S, Rosenblum M. The Baltimore Community-Based Organizations Neighborhood Network: Enhancing Capacity Together (CONNECT) Cluster RCT. Am J Prev Med. 2019 Aug;57(2):e31-e41. doi: 10.1016/j.amepre.2019.03.013. Epub 2019 Jun 25. PMID 31248746
- [Derived] Ibe CA, Basu L, Gooden R, Syed SB, Dadwal V, Bone LR, Ephraim PL, Weston CM, Wu AW; Baltimore CONNECT Project Team. From Kisiizi to Baltimore: cultivating knowledge brokers to support global innovation for community engagement in healthcare. Global Health. 2018 Feb 9;14(1):19. doi: 10.1186/s12992-018-0339-8. PMID 29426345

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We used the IRS Master file of Tax Exempt Organizations to identify all non-profit organizations in our zip codes of interest, and the used the NTEE (National Taxonomy of Exempt Entities) Classification System to exclude organizations that were not involved in the direct delivery of health and human services to adults.
Units Other Than Participants: Community-based Organizations
Groups:
- Intervention: This group was exposed to a multi-component intervention, which included: 1) Participation in monthly meetings with other Community Organization partners, 2) a subscription to a web-based platform called 'Healthify' ("a platform used by care teams to make quick and accurate referrals for patients who need additional help from social services", 3) provision of a Research Assistant to volunteer at the organization and to provide technical assistance with the use of Healthify, 4) access to a website with Health Education materials for patients provided in English and Spanish, information about recruiting volunteers, and information about upcoming professional training, and 5) participation in Meet and Greet Sessions with Johns Hopkins Health System inpatient and outpatient Social Workers and Case Managers.
- Control: This group did not participate in any intervention activities.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 2637; 11 Community-based Organizations | 4130; 11 Community-based Organizations
Completed | 2637; 10 Community-based Organizations | 4130; 10 Community-based Organizations
Not Completed | 0; 1 Community-based Organizations | 0; 1 Community-based Organizations

BASELINE CHARACTERISTICS:
Population: The baseline characteristics describe demographic information about the J-CHiP patients who were each assigned to a 'proximal' CBO from the twenty participating. The average utilization outcomes and changes among the patients assigned to each of the CBOs constituted the CBO-level outcomes for the primary analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention CBOs | Control CBOs | Total
Number analyzed (Participants) | 2637 | 4130 | 6767
Age, Continuous [Median (Full Range); unit: years] | 62 [12 to 89] | 62 [18 to 89] | 62 [12 to 89]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 1685 | 2584 | 4269
  Gender: Male | 951 | 1545 | 2496
  Gender: Unknown | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: African American | 1441 | 2089 | 3530
  Race/Ethnicity: Asian | 22 | 26 | 48
  Race/Ethnicity: Caucasian | 968 | 1704 | 2672
  Race/Ethnicity: Hispanic | 15 | 21 | 36
  Race/Ethnicity: Native American | 1 | 10 | 11
  Race/Ethnicity: Other | 114 | 167 | 281
  Race/Ethnicity: Unknown | 76 | 113 | 189
Insurance Type [Count of Participants; unit: Participants]
  Medicare | 1699 | 2664 | 4363
  PPMCO | 938 | 1466 | 2404

OUTCOME MEASURES:

1. Primary Outcome: Change in Emergency Department Visits + Hospital Days
Description: The change in the average number of monthly emergency department visits and days spent in the hospital from the pre- intervention to the post-intervention period for J-CHiP patients assigned to each of the CBOs, adjusted for baseline prognostic variables.
Time Frame: Pre-Intervention (09/01/2012 to 03/09/2014); Post-Intervention (03/10/2014-09/30/2015
Population: Data collected at the community-based organization level.
Measure: Mean (Standard Deviation); unit: Diff in monthly hospital days+ED visits
Units Other Than Participants: community based organizations
Groups:
- Control CBOs: For each of the 10 CBOs randomized to the control arm, we calculated the average change (adjusted for pre-intervention variables) from the pre-intervention (9/1/12 to 3/9/14) to the post-intervention post-intervention (3/10/14 to 9/30/15) periods in the monthly average of the number of ED visits and days spent in the hospital among all J-CHiP patients assigned to that arm.
- Intervention CBOs: For each of the 10 CBOs randomized to the intervention arm, we calculated the average change (adjusted for pre-intervention variables) from the pre-intervention (9/1/12 to 3/9/14) to the post-intervention post-intervention (3/10/14 to 9/30/15) periods in the monthly average of the number of ED visits and days spent in the hospital among all J-CHiP patients assigned to that arm.
Arm/Group | Control CBOs | Intervention CBOs
Number analyzed (Participants) | NA | NA
Number analyzed (community based organizations) | 10 | 10
Diff in monthly hospital days+ED visits | -0.0069 (0.513) | 0.0113 (0.525)
Statistical Analysis 1: Comparison: Control CBOs vs Intervention CBOs; The difference between the average sum of the number of days spent in the hospital and ED visits in the past month, pre- and post-intervention, adjusted for pre- intervention variables, was calculated for each patients. The average change scores among patients assigned to each CBO defined the CBO-level outcomes. We calculated a weighted average of the CBO outcomes separately for the iCBOs and cCBOs, defining the difference-in-differences statistic as the difference between the two averages; Test type: Other — The significance of the difference-in-differences statistic was assessed using randomization inference, a non-parametric permutation test. Confidence intervals were determined by inversion of the test statistic; p = 0.63, Randomization inference — We calculated the proportion of permuted statistics with values higher in magnitude than that of the observed adjusted difference in differences (the p-value). We inverted the test statistic to determine confidence intervals; Difference in differences = 0.0182, 95% CI 2-sided [-0.12 to 0.11] — The estimation parameter is the difference between the average adjusted change in the monthly ED visits and hospital days from the pre- to post- intervention periods for the patients assigned to the iCBOs as compared to the cCBOs

ADVERSE EVENTS:
Description: Adverse events data not collected.
Groups:
- Intervention: Proximity to an intervention community based organization (CBO)
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes